CLINICAL TRIAL: NCT07033039
Title: Effects of Photobiomodulation With Red and Infrared Low-level Laser Diodes in Individuals Undergoing Rhinoplasty at a Single Centre: Protocol for a Randomized, Double-blind, Controlled Clinical Trial
Brief Title: Effects of Red and Infrared Photobiomodulation in Rhinoplasty at a Single Centre
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Cinthya Cosme Gutierrez Duran, PhD, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 7.503.097
Record Dates: First submitted 2025-06-13; First posted 2025-06-24 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Rhinoplasty; Edema
Keywords: Photobiomodulation; Low-Level Laser Therapy; Postoperative; Inflammation
MeSH Terms: conditions — Edema; Inflammation | interventions — Low-Level Light Therapy

STUDY DESIGN:
Intervention Model Description: randomized, controlled, single centre, double-blind clinical trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Only the researcher responsible for administering the treatments, who will open the randomization envelopes, will be aware of the participants' group allocation. Group identification will be disclosed only after statistical analysis, ensuring blinding of all other individuals involved in the study.
  The researcher responsible for data collection, including the assessment of edema and all secondary outcomes, as well as the statistician, will remain blinded to group assignments. Additionally, participants will not be informed of the intervention received.
  To ensure blinding, the device will remain turned off for the control group, and its use will be simulated by the healthcare professional responsible for administering the photobiomodulation (PBM). The device sound will also be reproduced to simulate activation, ensuring that participants are unaware of differences between interventions.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Photobiomodulation Group (Experimental): Participants will receive active photobiomodulation (PBM) one hour before rhinoplasty, in addition to standard surgical and perioperative care.
  Interventions: Device: Photobiomodulation; Procedure: Standard treatment protocol
- Simulation of Photobiomodulation Group (Sham Comparator): Participants will receive a sham photobiomodulation procedure one hour before rhinoplasty, in addition to standard surgical and perioperative care.
  Interventions: Other: Simulation of Photobiomodulation; Procedure: Standard treatment protocol

INTERVENTIONS:
Device: Photobiomodulation — The photobiomodulation device used in this study will be the ECCO Reability (Ecco Fibras, Campinas, SP, Brazil), which is approved for clinical use by the Brazilian Health Regulatory Agency (ANVISA) under registration number 80323310001. The equipment is also certified by INMETRO, ensuring adherence to nationally established safety and performance standards.
  Arms: Photobiomodulation Group
Other: Simulation of Photobiomodulation — In the sham group, the photobiomodulation procedure will be simulated with the device turned off. To preserve blinding, the equipment will be positioned as in the active treatment and its operational sound will be reproduced during the simulation, ensuring that the intervention remains indistinguishable from the actual PBM application.
  Arms: Simulation of Photobiomodulation Group
Procedure: Standard treatment protocol — All participants will undergo primary open rhinoplasty performed using piezo-assisted osteotomies, following standardized surgical protocols. Subperiosteal dissection will be carried out along the lateral nasal walls, with supraperiosteal dissection in the medial region of the bony nasal dorsum. The configuration of osteotomies will be selected according to individual anatomical and surgical requirements. All procedures will be performed by experienced otolaryngologists.
  All participants will also receive standardized perioperative medical care, identical in both groups. No medication will be administered preoperatively. Intraoperatively, dexamethasone 4 mg and tranexamic acid 1 g will be administered intravenously. Postoperative in-hospital care will include hydrocortisone 200 mg IV, tranexamic acid 250 mg IV, dipyrone 1 g IV, and cefazolin 1 g IV every 8 hours, with ketorolac 10 mg sublingual as needed. After discharge, patients will receive cefuroxime axetil 500 mg orally every 12

SUMMARY:
This single-centre, randomized, double-blind, controlled clinical trial aims to evaluate the effectiveness of preoperative photobiomodulation (PBM) with red and infrared wavelengths in reducing periorbital edema in patients undergoing rhinoplasty. Sixty participants will be randomized to receive either active PBM or sham PBM one hour before surgery. The primary outcome is periorbital edema on postoperative day 3, assessed using the Hoffmann clinical scale, with standardized photographic analysis using ImageJ as a complementary measure. Secondary outcomes include the time course of periorbital edema, periorbital ecchymosis, postoperative pain, nasal tip skin thickness, analgesic consumption, and patient-reported functional and aesthetic outcomes assessed with the Standardized Cosmesis and Health Nasal Outcomes Survey (SCHNOS). Participants will be followed for up to 12 months postoperatively

DETAILED DESCRIPTION:
Edema and ecchymosis are common sequelae after rhinoplasty and may delay postoperative recovery and negatively affect patient satisfaction. These manifestations are related to the inflammatory cascade triggered by surgical trauma, leading to increased vascular permeability and tissue swelling. Photobiomodulation (PBM) is a non-invasive intervention that uses low-level light to modulate biological processes, including inflammation, pain, and tissue repair, and has demonstrated beneficial effects in several clinical contexts. However, evidence regarding its effectiveness in rhinoplasty remains limited.

This study is a single-centre, randomized, double-blind, controlled clinical trial designed to evaluate the effectiveness of preoperative PBM in reducing periorbital edema after rhinoplasty. A total of 60 participants undergoing primary open rhinoplasty with piezo-assisted osteotomies will be randomly allocated in a 1:1 ratio to either an experimental group or a control group. Participants in the experimental group will receive active PBM, while those in the control group will receive a sham PBM procedure. Both interventions will be applied one hour before surgery.

Photobiomodulation will be administered one hour before surgery by a trained healthcare professional using a standardized protocol with red and infrared wavelengths. In the control group, a sham procedure will be performed with the device turned off, with simulation of the procedure to maintain blinding. All participants will receive identical standardized surgical techniques and perioperative pharmacological care, which are not considered part of the study intervention.

The primary outcome of the study is periorbital edema on postoperative day 3, assessed using the Hoffmann clinical ordinal scale (0-4) by a calibrated assessor blinded to group allocation. Standardized photographic documentation analyzed with ImageJ software will be used as a complementary objective measure. Secondary outcomes include the time course of periorbital edema, periorbital ecchymosis, postoperative pain assessed using a visual analog scale, nasal tip skin thickness, analgesic consumption, and patient-reported functional and aesthetic outcomes assessed using the Standardized Cosmesis and Health Nasal Outcomes Survey (SCHNOS). Follow-up assessments will be conducted for up to 12 months after surgery.

Statistical analyses will be performed according to data distribution. The primary analysis will consist of a between-group comparison of periorbital edema on postoperative day 3, assessed using an ordinal clinical scale, and will therefore be conducted using non-parametric methods. Secondary outcomes will be analyzed descriptively and inferentially, as appropriate. All analyses will follow a modified intention-to-treat approach, including all randomized participants with at least one postoperative assessment. A two-sided significance level of 0.05 will be adopted. No interim analyses are planned. Adverse events will be monitored throughout the study period and reported in accordance with ethical and regulatory requirements

ELIGIBILITY:
Inclusion Criteria

* Age 18 to 60 years
* ASA physical status I or II
* No comorbidities (no pre-existing diseases)
* Scheduled for primary open rhinoplasty with piezo-assisted osteotomies
* Able and willing to provide written informed consent Exclusion Criteria
* Indication for secondary or revision rhinoplasty
* Indication for closed rhinoplasty
* Procedures not performed using piezo-assisted osteotomies
* Intraoperative complications (e.g., haemorrhage or technical difficulties)
* Use of anticoagulant, anti-inflammatory, or corticosteroid medications
* Prior nasal filler with hyaluronic acid
* Use of vitamin A derivatives (oral isotretinoin or topical retinoic acid) within 30 days before surgery
* Known allergy to any mandatory intra- or postoperative medication

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01-30 (Actual); Primary Completion 2029-11-30 (Estimated); Study Completion 2030-11-30 (Estimated)

PRIMARY OUTCOMES:
Periorbital Edema on postoperative day 3 | Postoperative day 3
  Periorbital edema assessed on postoperative day 3 using the Hoffmann clinical scale (0-4), based on eyelid involvement, evaluated by a blinded and calibrated assessor. Standardized photographic analysis using ImageJ will be used as a complementary objective measure.

SECONDARY OUTCOMES:
Periorbital Edema Time Course | 7, 30, 60, and 90 days; 6 and 12 months postoperatively
  Periorbital edema assessed using the Hoffmann clinical scale (0-4), based on eyelid involvement, evaluated by a blinded and calibrated assessor, with standardized photographic documentation and complementary ImageJ analysis.
Periorbital Ecchymosis | 3, 7, 30, 60, and 90 days; 6 and 12 months postoperatively
  Periorbital ecchymosis assessed using the Hoffmann clinical ordinal scale (0-4), based on the extent and intensity of periorbital discoloration, evaluated by a trained assessor blinded to group allocation.
Nasal Tip Skin Thickness | Preoperative baseline; 3, 7, 30, 60, and 90 days; 6 and 12 months postoperatively
  Skin thickness will be assessed through physical examination of the nasal tip using a standardized protocol. The evaluations will be conducted by a trained clinician during scheduled follow-up visits.
Postoperative Pain (VAS) | 3 and 7 days postoperatively
  Postoperative pain will be assessed using the Visual Analog Scale (VAS), a validated tool commonly used in rhinoplasty research. A 10 cm horizontal ruler will be used, with endpoints labeled "0" (no pain) and "10" (worst imaginable pain),. All participants will use the same standardized ruler.
Patient-Reported Functional and Aesthetic Outcomes (SCHNOS) | Preoperative baseline; 30 and 90 days; 6 and 12 months postoperatively
  Functional and aesthetic outcomes assessed using the Standardized Cosmesis and Health Nasal Outcomes Survey (SCHNOS), validated for Brazilian Portuguese.
Analgesic Consumption | 3, 7, 30, 60, and 90 days; 6 and 12 months postoperatively
  Total amount of analgesic medication ingested by each participant, recorded as an indirect indicator of postoperative pain control and functional recovery.

CONTACTS AND LOCATIONS:
Overall Officials: Cinthya CG Duran, PhD, Principal Investigator — University of Nove de Julho
Locations (1):
- Hospital Paulista de Otorrinolaringologia, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol